CLINICAL TRIAL: NCT02596308
Title: Immunogenicity and Safety of Subunit Plague Vaccine Comprised by Fraction 1 Capsule (F1) and Virulence-Associated (V) Antigens: A Random Phase 2a Clinical Trial
Brief Title: Immunogenicity and Safety of Subunit Plague Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Lanzhou Institute of Biological Products Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT017
Record Dates: First submitted 2015-11-02; First posted 2015-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Plague
Keywords: Plague vaccine; Immunogenicity; Safety
MeSH Terms: conditions — Plague | interventions — Plague Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 15µg vaccine (Experimental): 15µg plague vaccine of 1.0ml in 120 adults aged 18-55 years old at day 0 and 28.
  Interventions: Biological: Plague vaccine
- 30µg vaccine (Experimental): 30µg plague vaccine of 1.0ml in 120 adults aged 18-55 years old at day 0 and 28.
  Interventions: Biological: Plague vaccine

INTERVENTIONS:
Biological: Plague vaccine — Plague vaccine is comrised by native fraction 1 capsule (F1) and recombine virulence-associated (V) antigens.

SUMMARY:
Plague is a potentially fatal infection in humans caused by the bacterium Yersinia pestis. Pneumonic plague is typically diagnosed in humans with high mortality. It has a long history for plague as an agent of biowarfare, and poses a serious threat to international security. Althought the killed whole-cell plague vaccine and live attenuated vaccine have been licensed, they are rarely used today because of toxicities, limited evidence for efficacy to prevent plague, and limited commercial availability. In the last twenty years,the recombinant subunit vaccines comprised by fraction 1 capsule(F1)and virulence-associated (V)antigens as the main composition have caused widely attention with providing greater protection than vaccines comprised of either subunit alone. This study was aimed to explor the safety and immunogenicity of a new type plague subunit vaccine which comprised natural F1 antigen and recombined V antigen (F1+rV).

DETAILED DESCRIPTION:
Plague is a potentially fatal infection in humans caused by the bacterium Yersinia pestis, transmitted naturally from rodent reservoirs to humans via fleas. Human diseases may also result from contact with blood or tissues of infected animals or exposure to aerosolized droplets containing bacteria. Pneumonic plague is typically diagnosed in humans with with high mortality. It has a long history for plague as an agent of biowarfare, and poses a serious threat to international security. In human history, there were three outbreaks of plague all over the world, about 200 million people died from the disease. The increasing trend of plague epidemic in recent years, some regions and countries in the world still have the outbreak of the plague. It implies that safe and effective vaccine is urgently to developing. Althought the killed whole-cell plague vaccine and live attenuated vaccine have been licensed, these vaccines cause significant adverse reactions, including fever, headache, malaise, lymphadenopathy, erythema and induration at the injection site with high degree of immune variability. They are rarely used today because of toxicities, limited evidence for efficacy to prevent plague, and limited commercial availability. Based on the researches in the last twenty years,the recombinant subunit vaccines comprised by fraction 1 capsule(F1)and virulence-associated (V)antigens as the main composition have caused widely attention with providing greater protection than vaccines comprised of either subunit alone. This study was aim to exploring the safety and immunogenicity of a new type plague subunit vaccine which comprised by native F1 antigen and recombined V antigen (F1+rV).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-55months old as established by medical history and clinical examination.
* The subjects' guardians are able to understand and sign the informed consent.
* Subjects who can and will comply with the requirements of the protocol.
* Subjects with temperature ≤37.0°C on axillary setting.

Exclusion Criteria:

* Family history of seizures or progressive neurological disease.
* Subject who has a medical history of plague, or had been vaccination of plague vaccine.
* Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine.
* Any confirmed or suspected autoimmune diseases or immune deficiency disorders, including human immunodeficiency virus (HIV) infection.
* Dysgenopathy or severe chronic disease.
* Pregnant or lactating women.
* Women of reproductive age without contraception.
* Thrombocytopenia or other blood coagulation disorder, may cause taboo of intramuscular injection.
* Any prior administration of immunodepressant or corticosteroids, and antianaphylactic treatment, cytotoxic therapy in last 6 months.
* Difficult to collecting blood sample.
* Any prior administration of blood products in last 3 month.
* Any prior administration of other research medicines in last 1 month.
* Any prior administration of attenuated live vaccine in last 4 weeks.
* Any prior administration of subunit or inactivated vaccines in last 2 weeks.
* Had fever before vaccination, subjects with temperature >37.0°C on axillary setting.
* Rash on the injection site that may affect safety observation.
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives.

Exclusion Criteria for the second dose:

* Subject who must be excluded according to the exclusion criteria for the first dose.
* Any serious adverse events caused by vaccination.
* Hypersensitivity after vaccination (include urticarial or rash in 30 minutes after vaccination).Hypersensitivity after vaccination (include urticarial or rash in 30 minutes after vaccination).
* Other adverse reactions in the opinion of the investigator that affect continue vaccination (include: severely serious symptom of pain, swelling, Limitation of motion, continuous high fever, headache and other Systemic or local reactions).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To evaluate immunogenicity after vaccination. | Day 28 post-dose 2
  the GMT of antibodies to F1 antigen at day 28 post-dose2
Proportion of subjects reporting solicited adverse reactions. | Day 7 post-each dose
  Proportion of subjects reporting solicited adverse events within 7 days post-each dose

SECONDARY OUTCOMES:
GMI of antibodies to F1 antigen. | Day 28 post-each dose
The seroconversion rate of antibodies to F1 antigen | Day 28 post-each dose
GMT of antibodies to F1 antigen at day 28 | Day 28 post- dose1
GMT of antibodies to V antigen. | Day 28 post-each dose
GMI of antibodies to V antigen. | Day 28 post-each dose
The seroconversion rate of antibodies to V antigen. | Day 28 post-each dose
Proportion of subjects reporting unsolicited adverse events | Day 28 post-each dose
  Proportion of subjects reporting unsolicited adverse events within 28 days post-each dose
Proportion of subjects with serious adverse events (SAE)occurring throughout the trial | Day 0 up to day 28 post-dose 2
  Proportion of subjects with serious adverse events (SAE)occurring throughout the trial from day 0 to 56.

CONTACTS AND LOCATIONS:
Overall Officials: Yuemei Hu, Bachelor, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Hu J, Jiao L, Hu Y, Chu K, Li J, Zhu F, Li T, Wu Z, Wei D, Meng F, Wang B. One year immunogenicity and safety of subunit plague vaccine in Chinese healthy adults: An extended open-label study. Hum Vaccin Immunother. 2018;14(11):2701-2705. doi: 10.1080/21645515.2018.1486154. Epub 2018 Jul 11. PMID 29927704